CLINICAL TRIAL: NCT00373607
Title: Phase 3a: Efficacy, Safety, and Tolerability of Dihydroartemisinin/Piperaquine (Artekin®) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Peruvian Amazon Region
Brief Title: Efficacy and Safety of Dihydroartemisinin/Piperaquine (Artekin®) for the Treatment of Uncomplicated Malaria in Peru
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: prof Umberto D'Aessandro, Institute of Tropical Medicine, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTEKINPERU
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Malaria
Keywords: Non complicated malaria; Microscopy; Adult; Children
MeSH Terms: conditions — Malaria | interventions — Mefloquine; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dihydroartemisin-piperaquine (Experimental): Dihydroartemisin-piperaquine (Artekin, Hualijian Pharmaceutical Co. Ltd., Guangzhou, China). Each tablet contains 40mg of dihydroartemisinin and 320mg piperaquine
  Interventions: Drug: Dihydroartemisin-piperaquine
- Mefloquine + Artesunate (MAS3) (Active Comparator): The MAS3 regimen is artesunate 4 mg/kg/day once daily for 3 days plus mefloquine 24 mg/kg given as a three day regimen of 8mg/kg/day
  Interventions: Drug: Mefloquine + Artesunate

INTERVENTIONS:
Drug: Dihydroartemisin-piperaquine — Dihydroartemisin-piperaquine (Artekin) manufactured by Hualijian Pharmaceutical Co. Ltd., Guangzhou, China. Each tablet contains 40mg of dihydroartemisinin and 320mg piperaquine
  Other Names: Artekin
  Arms: Dihydroartemisin-piperaquine
Drug: Mefloquine + Artesunate — Mefloquine + Artesunate (MAS3). The regimen is artesunate 4 mg/kg/day once daily for 3 days plus mefloquine 24 mg/kg given as a three day regimen of 8mg/kg/day
  Other Names: MAS3
  Arms: Mefloquine + Artesunate (MAS3)

SUMMARY:
In Peru, Mefloquine plus Artesunate (MAS3), is the current first line treatment for P. falciparum malaria in the Amazonian Region, and has proved its efficacy against multi-resistant P. falciparum parasites, but several side effects have been reported. Dihydroartemisinin-piperaquine (DHA-PPQ) is a new co-formulated and well tolerated ACT, increasingly used in Southeast Asia where it has proved to be highly effective against Plasmodium falciparum malaria. We tested the efficacy, safety and tolerability of DHA-PPQ in patients with uncomplicated P. falciparum malaria. A RCT to evaluate DHA-PPQ was carried out, between 2003 and 2005. Patients with uncomplicated P. falciparum malaria were randomly allocated to receive either DHA-PPQ or MAS3 with a 63-day follow-up period. Five hundred twenty two patients were included in the analysis, 262 were allocated to receive DHA-PPQ, and 260 to receive MAS3. The two groups were comparable at baseline in demographic and clinical characteristics. The mean time for parasite clearance into the DHA-PPQ group was 32.0 hours and 35.5 hours in the MAS3 group. Twenty-four hours after the first dose, the proportions of patients whose cleared parasitaemia were 67.2% in the DHA-PPQ group, and 58.1% in the MAS3 group (RR 1.25, [95% CI 1.03-1.52], p = 0.017). All patients were able to clear parasites within 72 hours after the first dose. The mean time for fever clearance was 28.0 and 29.5 hours in DHA-PPQ and MAS3 group respectively. (P= 0.69). Twenty-four hours after the first dose, 85.5% and 83.1% of patients cleared fever in the DHA-PPQ and MAS3 group respectively (p>0.05). The Adequate Clinical and Parasitological Response (ACPR), PCR adjusted, were 97.7% and 99,2% for the DHA-PPQ and MAS3 group respectively, (RR 0.99, 95% CI [0.86-1.13], P = 0.88). No Early Treatments Failures were reported in any group. In the DHA-PPQ group, according to the PCR adjusted results, 6 subjects had Late treatment Failures. In the MAS3 group, two Late Treatment Failures was reported. The frequency of adverse events was significantly lower in patients treated with DHA-PPQ than in those treated with MAS3.

DHA-PPQ proved to be a highly effective antimalarial drug for the treatment of P. falciparum malaria and suitable for use in the Peruvian Amazon region. It also has the advantage of being better tolerated. In terms of cost, DHA-PPQ is cheaper and more affordable than MAS3 and should be considered for the National Antimalarial Drug Policy in Perú.

DETAILED DESCRIPTION:
In Peru, Mefloquine plus Artesunate (MAS3), is the current first line treatment for P. falciparum malaria in the Amazonian Region, and has proved its efficacy against multi-resistant P. falciparum parasites, but several side effects have been reported. Dihydroartemisinin-piperaquine (DHA-PPQ) is a new co-formulated and well tolerated ACT, increasingly used in Southeast Asia where it has proved to be highly effective against Plasmodium falciparum malaria. We tested the efficacy, safety and tolerability of DHA-PPQ in patients with uncomplicated P. falciparum malaria. A RCT to evaluate DHA-PPQ was carried out, between 2003 and 2005. Patients with uncomplicated P. falciparum malaria were randomly allocated to receive either DHA-PPQ or MAS3 with a 63-day follow-up period. Five hundred twenty two patients were included in the analysis, 262 were allocated to receive DHA-PPQ, and 260 to receive MAS3. The two groups were comparable at baseline in demographic and clinical characteristics. The mean time for parasite clearance into the DHA-PPQ group was 32.0 hours and 35.5 hours in the MAS3 group. Twenty-four hours after the first dose, the proportions of patients whose cleared parasitaemia were 67.2% in the DHA-PPQ group, and 58.1% in the MAS3 group (RR 1.25, [95% CI 1.03-1.52], p = 0.017). All patients were able to clear parasites within 72 hours after the first dose. The mean time for fever clearance was 28.0 and 29.5 hours in DHA-PPQ and MAS3 group respectively. (P= 0.69). Twenty-four hours after the first dose, 85.5% and 83.1% of patients cleared fever in the DHA-PPQ and MAS3 group respectively (p>0.05). The Adequate Clinical and Parasitological Response (ACPR), PCR adjusted, were 97.7% and 99,2% for the DHA-PPQ and MAS3 group respectively, (RR 0.99, 95% CI [0.86-1.13], P = 0.88). No Early Treatments Failures were reported in any group. In the DHA-PPQ group, according to the PCR adjusted results, 6 subjects had Late treatment Failures. In the MAS3 group, two Late Treatment Failures was reported. The frequency of adverse events was significantly lower in patients treated with DHA-PPQ than in those treated with MAS3.

DHA-PPQ proved to be a highly effective antimalarial drug for the treatment of P. falciparum malaria and suitable for use in the Peruvian Amazon region. It also has the advantage of being better tolerated. In terms of cost, DHA-PPQ is cheaper and more affordable than MAS3 and should be considered for the National Antimalarial Drug Policy in Perú.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5 - 60 years old
* Fever (axillary temperature equal or higher than 37,5 °C) or history of fever in the previous 24 hours
* Monoinfection with P. falciparum, with parasitic density between 1,000 and 200,000 par/µl
* Informed consent provided by patient or parent or legal tutor

  • Exclusion criteria:
* Mixed malaria infection
* Pregnancy or breastfeeding to child ≤ 6 months of age
* One or more danger signs or any sign of severe or complicated malaria
* A concomitant severe disease
* History of treatment with mefloquine in the last 60 days or chloroquine, primaquine or quinine within the 14 days before the present episode
* History of neuropsychiatric disease
* History of hypersensitivity reactions to artemisinins or mefloquine
* History of splenectomy

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 522 (Actual)
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Adequate Clinical and parasitological response | Day 63

SECONDARY OUTCOMES:
Recrudescence | Day 63
Reinfections | day 63
SAE | Day 63
AE | Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD,MSc, PHD, Study Director — Institute of Tropical Medicine Antwerp

REFERENCES:
- [Derived] Grande T, Bernasconi A, Erhart A, Gamboa D, Casapia M, Delgado C, Torres K, Fanello C, Llanos-Cuentas A, D'Alessandro U. A randomised controlled trial to assess the efficacy of dihydroartemisinin-piperaquine for the treatment of uncomplicated falciparum malaria in Peru. PLoS One. 2007 Oct 31;2(10):e1101. doi: 10.1371/journal.pone.0001101. PMID 17971864